CLINICAL TRIAL: NCT05926154
Title: Evaluation of Ischemia and Reperfusion Interval With Neuromonitorization in Tourniquet Application
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, AHMET MUCTEBA YILDIRIM, Principal Investigator, MD, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: Low Extremity neuromonitoring
Record Dates: First submitted 2023-05-07; First posted 2023-07-03 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Quadriceps Muscle Atrophy; Tourniquet; EMG

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LOP + 50 mmHg (Experimental): As a result of randomization, the surgical tourniquet pressure is 50 mmHg higher than the limb occlusion pressure. Limb occlusion pressure is calculated using the formulation by Graham: LOP = [(Systolic Pressure - Diastolic Pressure)× (Limb Diameter) / 3 Cuff Width)] + Diastolic Pressure
  Interventions: Procedure: Surgical tourniquet pressure selection
- LOP + 100 mmHg (Experimental): As a result of randomization, the surgical tourniquet pressure is 100 mmHg higher than the limb occlusion pressure. Limb occlusion pressure is calculated using the formulation by Graham: LOP = [(Systolic Pressure - Diastolic Pressure)× (Limb Diameter) / 3 Cuff Width)] + Diastolic Pressure
  Interventions: Procedure: Surgical tourniquet pressure selection

INTERVENTIONS:
Procedure: Surgical tourniquet pressure selection — Limb occlusion pressure is calculated using the formulation by Graham: LOP = [(Systolic Pressure - Diastolic Pressure)× (Limb Diameter) / 3 Cuff Width)] + Diastolic Pressure. One group is LOP + 50 mm Hg and other one is LOP + 100 mmHg

SUMMARY:
The goal of this clinical trial is to compare two differential tourniquet pressure in lower extremity surgery cases. The main questions it aims to answer are:

* What are the perioperative neurophysiological effects of ischemia and compression in the tissue under the tourniquet?
* Are the effects of two different tourniquet pressures on neuromonitoring significantly different?
* Can the ideal time of the reperfusion interval be evaluated by neuromonitoring?
* Are the effects of two different tourniquet pressures on the quadriceps denervation significantly different from each other? Participants meeting the inclusion criteria will be evaluated for parameters to be used preoperatively. It will be evaluated in the 1st day, 1st week and 1-month follow-ups in the postoperative period.

The investigators will compare two different tourniquet pressure ( Limb occlusion pressure +50 mmHg / + 100 mmHg) to see if it will be evaluated whether there is a significant difference in terms of quadriceps denervation, vas scores, total blood estimate volume loss, intraoperative MEP decrease, and recovery times, quadriceps tendon thickness, thigh circumfrences.

DETAILED DESCRIPTION:
As a result of the power analysis for this study, the number of samples was determined as 24. The study was started after the approval of the ethics committee.

Participants who met the inclusion and exclusion criteria were randomized in terms of tourniquet pressure to be applied and divided into two groups. It was planned to evaluate quadriceps tendon thickness by USG and MRI, thigh circumference, VAS scores, CBC, and CK in blood samples in the preoperative period of all patients. It was planned to obtain parameters related to MEP by using intraoperative neuromonitorization during the surgery. In the postoperative period, all parameters that were evaluated preoperatively on the 1st day, 1st week, and 1st month were re-evaluated. Finally, EMG evaluation was planned for 1 month.

ELIGIBILITY:
Inclusion Criteria:

* Operation planning in the foot and ankle area

Exclusion Criteria:

* Having a history of previous foot and ankle surgery,
* Having a history of previous knee surgery or spinal surgery,
* Diagnosis of diabetes mellitus,
* Having a known diagnosis of a disease affecting the peripheral nervous system (peripheral neuropathy, previous spinal surgery, stroke, etc.),
* Having a diagnosis of a disease affecting the known peripheral vascular system (Peripheral vascular disease, calcified popliteal artery, peripheral arterial bypass surgery, vasculitis, advanced chronic venous insufficiency),
* Having a disease that affects the ideal tourniquet application (Chronic Lymphedema, BMI>35, Stage 3 and above chronic renal failure, uncontrollable hypertension),
* Having been diagnosed with a known coagulation disorder,
* History of pulmonary embolism or deep vein thrombosis.
* ASA score above 3
* Surgery time to be less than 80 minutes

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-11 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
MEP 50% reduction in intraoperative neuromonitorization | Intraoperative
  Time with more than 50% reduction in perioperative MEP will be compared in groups in which two different tourniquet pressures were applied.
MEP full recovery intraoperative neuromonitorization | Intraoperative
  Time with full recovery in perioperative MEP will be compared in groups in which two different tourniquet pressures were applied.

SECONDARY OUTCOMES:
Quadriceps Tendon Thickness-USG | Preoperative, Postoperative 1st day and 4th week will be evaluated
  In the study, quadriceps tendon thickness measurements will be performed in B Mode using the Clarius Portable L7 HD3 Linear Ultrasound device (13-4 MHz).The measurements of the patients will be performed in the supine position with the knee flexed to 30 degrees with a pillow placed in the popliteal web to prevent anisotropy in the quadriceps. The USG probe will be parallel to the long axis of the femur in the sagittal plane, and the patella will be placed at the midpoint of the proximal pole with its distal part. Quadiceps tendon thickness was measured at three different levels, 5-10-15 mm from the proximal patella. The quadriceps tendon borders were determined as the first hyperechoic region, superficial and deep.
Quadriceps Tendon Thickness-MRI | Preoperative, Postoperative third month
  In the study, the thickness of the quadriceps tendon will also be evaluated with MRI. In the sagittal T1 sequence of knee MRI images, the portion with the largest diameter 1.5 and 3 cm proximal to the superior pole of the patella will be taken as the tendon thickness.
Thigh Diameter | Preoperative, Postoperative 1st day, first week and 4th week will be evaluated
  Thigh diameters were measured comparatively with a non-flexible 7 mm tape measure from 10 cm proximal to the midpoint of the proximal patella. As the leg length, the distance from the level of the tibial plateau to the medial malleolus type was measured.
Total Blood Estimate Volume Loss | Preoperative, Postoperative 1st day
  Total blood volume will be calculated with the formula Nadler previously presented in the literature. Total blood volume loss will be calculated using preoperative and postoperative hemogram and hematocrit parameters.
CK levels | Preoperative, Postoperative 1st day, Postoperative 1 st month
  Creatinine kinase, one of the blood parameters showing muscle degradation, will be evaluated by taking blood samples from the patients before and after the surgery.
EMG | Postoperative 1 st month
  ENMG is an electrophysiological study often used to evaluate nerve injuries. Permanent nerve damage will be evaluated with a nerve conduction study performed by an experienced neurologist comparing both extremities at the first postoperative month of the participants. Peroneal and tibial nerves as motor nerves, sural and s.peroneal nerves as sensory nerves will be evaluated. The latency, amplitude and nerve conduction velocities of the nerves will be compared.
Surgical Area Pain | Preoperative, Postoperative 1st day, Postoperative 1 st month
  The pain of the surgical area will be evaluated over the VAS score.

CONTACTS AND LOCATIONS:
Overall Officials: Serkan BAYRAM, Ass. Prof., Study Director — Istanbul University Medicine Faculty Orthoapedic and Traumatology Department
Locations (1):
- Department of Orthopaedics and Traumatology, Istanbul University, Istanbul, Turkey, Istanbul, Fatih-Topkapı, Turkey (Türkiye)

REFERENCES:
- [Derived] Yildirim AM, Bayram S, Kizilkurt T, Canbolat N, Baslo MB, Asik M. Low tourniquet pressure has less impact on lower extremity nerve innervation: comparison of different tourniquet pressures used with intraoperative neuromonitoring with a randomized controlled study. J Orthop Surg Res. 2024 Oct 23;19(1):684. doi: 10.1186/s13018-024-05176-y. PMID 39444003